CLINICAL TRIAL: NCT04531189
Title: Clinical Evaluation and Assessment of Instruments and Biomarkers in Subjects With Wilson Disease
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX701-CL001
Record Dates: First submitted 2020-07-27; First posted 2020-08-28 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample for future UX701 related research (DNA, RNA, proteins)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to determine the relevance and appropriateness of outcome assessments, including biomarkers, within the Wilson disease population to inform study design and endpoint selection for future clinical studies.

DETAILED DESCRIPTION:
Given the limited information on the frequency and spectrum of disease manifestations and clinical course of Wilson disease, the UX701-CL001 study aims to assess the utility and feasibility of various assessments and biomarkers to inform endpoint selection for future clinical studies, better understand the relationship between biomarkers and potential clinical outcomes, and characterize the clinical presentation of Wilson disease. UX701-CL001 is a clinical survey study. Subjects will complete assessments at the study site and at home to evaluate the clinical manifestations of Wilson disease in clinical and real-world environments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age at the time written informed consent is provided.
2. Confirmed diagnosis of Wilson disease.
3. Have a documented history of copper chelator (ie, penicillamine, trientine) and/or zinc therapy or be ≥ 1 year post liver transplant with no active associated complications.
4. Willing and able to comply with all study procedures and requirements. If < 18 years of age (or as required by region), have a caregiver who is willing and able to assist with study requirements if needed.
5. Willing and able to provide written informed consent after the study has been explained and before any study-related data are collected or study-related procedures are performed. If < 18 years of age (or as required by region), willing and able to provide written assent and have a legally authorized representative who is willing and able to provide written informed consent after the study has been explained and before any study-related data are collected or study-related procedures are performed.

Exclusion Criteria:

1. History of liver disease due to a medical condition unrelated to Wilson disease.
2. Liver fibrosis stage F3 or F4.
3. Decompensated hepatic cirrhosis and/or evidence of portal hypertension.
4. Marked neurological disease requiring either nasogastric feeding or intensive inpatient medical care.
5. Female subject who is pregnant or breastfeeding or who plans to become pregnant at any time during the study.
6. Female subject of childbearing potential who has a positive urine pregnancy test on Day 1 or is unwilling to have additional pregnancy tests during the study.
7. Current or previous participation in a gene transfer study.
8. Presence or history of any disease or condition that, in the Investigator's opinion, would interfere with the subject's safety or ability to participate in the study or significantly affect interpretation of study results.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a confirmed diagnosis of Wilson Disease will be enrolled from outpatient clinics and metabolic genetic centers in the United States. Subjects may participate regardless of their current treatment. Subjects who have had a liver transplant for treatment of Wilson Disease are also invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Clinical manifestation of Wilson Disease under study: demographics | 30 days
Clinical manifestation of Wilson Disease under study: general medical history, Wilson Disease history and treatments | 30 days
Clinical manifestation of Wilson Disease under study: patient reported outcomes and clinician reported outcomes | 30 days
Clinical manifestation of Wilson Disease under study: activity monitoring | 30 days
Clinical manifestation of Wilson Disease under study: motor function | 30 days
Clinical manifestation of Wilson Disease under study: joint pain | 30 days
Clinical manifestation of Wilson Disease under study: serum copper biomarker assessments | 30 days
Clinical manifestation of Wilson Disease under study: 24-hour urinary copper concentration | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ultragenyx Medical Director, Study Director — Ultragenyx Pharmaceutical
Locations (6):
- United States (5):
  - Yale University School of Medicine, New Haven, Connecticut
  - Jackson Memorial Hospital Miami Transplant Unit University of Miami Miller School of Medicine, Miami, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Michigan Michigan Medicine Hepatology Clinic Taubman Center, Ann Arbor, Michigan
  - Seattle Children's Hospital, Seattle, Washington
- Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/Wilson Disease Information — https://ultrarareadvocacy.com/wilson-disease-wd/